CLINICAL TRIAL: NCT04651426
Title: Use of a Non-medicated Plaster in Chronic Lumbar Back Pain.
Acronym: CERFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Matteo Ricci, Associate Professor at Department of Orthopaedic Surgery, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2128CESC
Record Dates: First submitted 2020-10-17; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Back Pain
Keywords: non-medicated plaster, lumbar back pain, FIT Therapy
MeSH Terms: conditions — Back Pain; Low Back Pain

STUDY DESIGN:
Intervention Model Description: Prospective analysis in a 3-arm, randomized double-blind and placebo-controlled stud
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): The Placebo is a Patch identical to the F3 and F4 patches in aesthetics but without any biomineral, therefore with no reflectance ability.
  Interventions: Device: The FIT Therapy patch (D. FENSTEC s.r.l. Altavilla Vicentina, Italy) is a medical device class 1
- F3 Patch (Active Comparator): The F3 is a patch made of 100% polypropylene non-woven fabric, an acrylic adhesive mass and a mix of titanium dioxide printed on with a refringency spectrum 2 m x kg
  Interventions: Device: The FIT Therapy patch (D. FENSTEC s.r.l. Altavilla Vicentina, Italy) is a medical device class 1
- F4 Patch (Active Comparator): The F4 is a patch made of 100% polypropylene non-woven fabric, an acrylic adhesive mass and a mix of titanium dioxide printed on with a refringency spectrum of 4 m x kg
  Interventions: Device: The FIT Therapy patch (D. FENSTEC s.r.l. Altavilla Vicentina, Italy) is a medical device class 1

INTERVENTIONS:
Device: The FIT Therapy patch (D. FENSTEC s.r.l. Altavilla Vicentina, Italy) is a medical device class 1 — The FIT Therapy patch (D. FENSTEC s.r.l. Altavilla Vicentina, Italy) is a medical device class 1 which mechanism of action is through the ability of biominerals to reflect the far infrared radiation (FIR). Normally the human body temperature would dissipate regular far infrared radiations but, thanks to the FIT Therapy (Far Infrared Technology), these waves are reflected and allowed to reach deeper areas in the human body (wavelength spectrum is 4-21 µm with a denser concentration around 11 µm).
  Every FIT device act as a mirror and they are able to induce an antalgic effect simply thanks to this biophysical process, therefore without releasing any active ingredient or creating a thermic shock.
  The plasters are made of 100% polypropylene non-woven fabric, an acrylic adhesive mass and a mix of titanium dioxide printed on. This particular mix in powder form is characterized by particles sizes above 100 nm.

SUMMARY:
The investigator assessed 54 patients with chronic lumbar back pain treated with FIT Therapy (far infrared technology) patch. The criteria for inclusion were chronic lumbar back pain due to overstress or to contracture and patients over 30 years old. Patients with tumors, infections, neurological and metabolic diseases were excluded. Three different types of FIT Therapy patches (F4, F3 and the placebo) were used according to the different power of action. The patches were self-removed after 5 days. At day 8 new ones were applied for other five days and at day 14 patients were dismissed. Every single patient was assessed during the study using the VAS pain scale, the Roland Morris questionnaire for quality of life and the range of motion (ROM).

DETAILED DESCRIPTION:
First and foremost, the investigators obtained the ethical committee approval, then 54 patients were enrolled since May 2019 to November 2019, at the AOUI (Azienda Ospedaliera Universitaria Integrata) Verona. Prospective analysis in a 3-arm, randomized double-blind and placebo-controlled study was performed to assess the effect of FIT Therapy patches on the chronic lumbar spine pain and on the ROM.

The FIT Therapy patch (D. FENSTEC s.r.l. Altavilla Vicentina, Italy) is a medical device class 1 which mechanism of action is through the ability of biominerals to reflect the far infrared radiation (FIR).

Normally the human body temperature would dissipate regular far infrared radiations but, thanks to the FIT Therapy (Far Infrared Technology), these waves are reflected and allowed to reach deeper areas in the human body (wavelength spectrum is 4-21 µm with a denser concentration around 11 µm).

Every FIT device act as a mirror and they are able to induce an antalgic effect simply thanks to this biophysical process, therefore without releasing any active ingredient or creating a thermic shock.

The plasters are made of 100% polypropylene non-woven fabric, an acrylic adhesive mass and a mix of titanium dioxide printed on. This particular mix in powder form is characterized by particles sizes above 100 nm. The intrinsic properties of the FIT technology are due to the mix of titanium dioxides that reflect the FIR emitted by the human body.

Three different plasters were used: a placebo (without any biomineral, therefore with no reflectance ability); an "F3" patch and an "F4" one, characterized by different power of action (F4 has a broader spectrum of refrigency than F3). The 3 plasters presented no difference in size, color and shape.

Patients were subdivided in 3 randomized groups.The Visual Analogic Scale (VAS) and the Roland Morris Disability Questionnaire (RMDQ) were used. The Range of Motion (ROM) evaluation consisted of flexion and extension, lateral bending and rotation of the lumbar spine.

The trial consisted of a total of 14 days for each patient. At day 0, during the first clinical encounter, patients were enrolled by signing an informed consent. Still during the encounter, the lumbar spine ROM was measured, the VAS and the RMDQ administered. Only after all these necessary steps the first patch was applied. Every patient was given a RMDQ and a journal, which had to be updated daily, and at the same time every day, with the pain level experienced and any adverse effect to the FIT Therapy patch. At day 5 the patch was self-removed and the RMDQ given during the first encounter filled. The second clinical encounter was at day 8. The patients' ROM and VAS were tested for the second time and a new FIT Therapy patch was applied. At day 13 the FIT Therapy patch was dismissed and a second RMDQ filled at home. The last clinical encounter was held at day 14 and once again all 54 patients' ROM and VAS were assessed. Finally, the daily journal was collected, and patients were asked if any other pain medication was self-administered during the entirety of the tests.

ELIGIBILITY:
Inclusion Criteria::

* chronic lumbar spine pain due to muscle contractures or over-use
* a signed informed consent
* patients 30 years of age or older.

Exclusion Criteria:

* infections
* neoplastic masses
* neuropathies
* metabolic disorders triggering the lumbar pain

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
The changes induced by the different types of FIT Therapy patches (placebo, "F3" and "F4"), in the pain level due to lower back pain, measured on the VAS scale. | The VAS scale results were compared, between the different patches, at day 0, 5, 8 and 14.
  VAS scale (Visual Analogic Scale)

SECONDARY OUTCOMES:
Changes in the Range Of Motion (ROM) | The degrees of motion were absessed at day 0, day 8 and day 14
  Degrees of flexion-extension and lateral bending of the patient.

OTHER OUTCOMES:
Changes in lifestyle. | The results of the RMDQ were absessed at day 0, day 8 and day 14
  Evaluated on the median values of the RMDQ (Roland Morris Disability Questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Ricci, Professor, Principal Investigator — Azienda Ospedaliera Universitaria Integrata Verona
Locations (1):
- Azienda Ospedaliera Universitaria Integrata, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wong CH, Lin LC, Lee HH, Liu CF. The analgesic effect of thermal therapy after total knee arthroplasty. J Altern Complement Med. 2012 Feb;18(2):175-9. doi: 10.1089/acm.2010.0815. PMID 22339105
- [Background] Lee CH, Roh JW, Lim CY, Hong JH, Lee JK, Min EG. A multicenter, randomized, double-blind, placebo-controlled trial evaluating the efficacy and safety of a far infrared-emitting sericite belt in patients with primary dysmenorrhea. Complement Ther Med. 2011 Aug;19(4):187-93. doi: 10.1016/j.ctim.2011.06.004. Epub 2011 Jul 16. PMID 21827932
- [Background] Allegri M, Montella S, Salici F, Valente A, Marchesini M, Compagnone C, Baciarello M, Manferdini ME, Fanelli G. Mechanisms of low back pain: a guide for diagnosis and therapy. F1000Res. 2016 Jun 28;5:F1000 Faculty Rev-1530. doi: 10.12688/f1000research.8105.2. eCollection 2016. PMID 27408698
- [Background] Bagnato GL, Miceli G, Atteritano M, Marino N, Bagnato GF. Far infrared emitting plaster in knee osteoarthritis: a single blinded, randomised clinical trial. Reumatismo. 2012 Dec 20;64(6):388-94. doi: 10.4081/reumatismo.2012.388. PMID 23285483
- [Background] Lai CH, Leung TK, Peng CW, Chang KH, Lai MJ, Lai WF, Chen SC. Effects of far-infrared irradiation on myofascial neck pain: a randomized, double-blind, placebo-controlled pilot study. J Altern Complement Med. 2014 Feb;20(2):123-9. doi: 10.1089/acm.2013.0122. Epub 2013 Oct 23. PMID 24152215
- [Background] Ricci M, Micheloni GM, Perusi F, Corbo VR, Vecchini E, Magnan B. Use of a non-medicated plaster in shoulder tendinopathies. Acta Biomed. 2016 Apr 15;87 Suppl 1:90-4. PMID 27104326
- [Background] Hoy D, Bain C, Williams G, March L, Brooks P, Blyth F, Woolf A, Vos T, Buchbinder R. A systematic review of the global prevalence of low back pain. Arthritis Rheum. 2012 Jun;64(6):2028-37. doi: 10.1002/art.34347. Epub 2012 Jan 9. PMID 22231424
- [Background] Ma K, Zhuang ZG, Wang L, Liu XG, Lu LJ, Yang XQ, Lu Y, Fu ZJ, Song T, Huang D, Liu H, Huang YQ, Peng BG, Liu YQ. The Chinese Association for the Study of Pain (CASP): Consensus on the Assessment and Management of Chronic Nonspecific Low Back Pain. Pain Res Manag. 2019 Aug 15;2019:8957847. doi: 10.1155/2019/8957847. eCollection 2019. PMID 31511784
- [Background] Will JS, Bury DC, Miller JA. Mechanical Low Back Pain. Am Fam Physician. 2018 Oct 1;98(7):421-428. PMID 30252425
- [Background] Santos LF, Correia IJ, Silva AS, Mano JF. Biomaterials for drug delivery patches. Eur J Pharm Sci. 2018 Jun 15;118:49-66. doi: 10.1016/j.ejps.2018.03.020. Epub 2018 Mar 20. PMID 29572160
- [Background] Pastore MN, Kalia YN, Horstmann M, Roberts MS. Transdermal patches: history, development and pharmacology. Br J Pharmacol. 2015 May;172(9):2179-209. doi: 10.1111/bph.13059. Epub 2015 Mar 18. PMID 25560046
- [Background] Miller K. Transdermal patches: past, present and future. Ther Deliv. 2015;6(6):639-41. doi: 10.4155/tde.15.16. No abstract available. PMID 26149780
- [Background] Tsai SR, Hamblin MR. Biological effects and medical applications of infrared radiation. J Photochem Photobiol B. 2017 May;170:197-207. doi: 10.1016/j.jphotobiol.2017.04.014. Epub 2017 Apr 13. PMID 28441605
- [Background] Johnstone DM, Moro C, Stone J, Benabid AL, Mitrofanis J. Turning On Lights to Stop Neurodegeneration: The Potential of Near Infrared Light Therapy in Alzheimer's and Parkinson's Disease. Front Neurosci. 2016 Jan 11;9:500. doi: 10.3389/fnins.2015.00500. eCollection 2015. PMID 26793049
- [Background] Vatansever F, Hamblin MR. Far infrared radiation (FIR): its biological effects and medical applications. Photonics Lasers Med. 2012 Nov 1;4:255-266. doi: 10.1515/plm-2012-0034. PMID 23833705
- [Background] Oosterveld FG, Rasker JJ, Floors M, Landkroon R, van Rennes B, Zwijnenberg J, van de Laar MA, Koel GJ. Infrared sauna in patients with rheumatoid arthritis and ankylosing spondylitis. A pilot study showing good tolerance, short-term improvement of pain and stiffness, and a trend towards long-term beneficial effects. Clin Rheumatol. 2009 Jan;28(1):29-34. doi: 10.1007/s10067-008-0977-y. Epub 2008 Aug 7. PMID 18685882
- [Background] Hausswirth C, Louis J, Bieuzen F, Pournot H, Fournier J, Filliard JR, Brisswalter J. Effects of whole-body cryotherapy vs. far-infrared vs. passive modalities on recovery from exercise-induced muscle damage in highly-trained runners. PLoS One. 2011;6(12):e27749. doi: 10.1371/journal.pone.0027749. Epub 2011 Dec 7. PMID 22163272
- [Background] Yang X, Zhao X, Yang K, Liu Y, Liu Y, Fu W, Luo Y. Biomedical Applications of Terahertz Spectroscopy and Imaging. Trends Biotechnol. 2016 Oct;34(10):810-824. doi: 10.1016/j.tibtech.2016.04.008. PMID 27207226
- [Background] Romanenko S, Begley R, Harvey AR, Hool L, Wallace VP. The interaction between electromagnetic fields at megahertz, gigahertz and terahertz frequencies with cells, tissues and organisms: risks and potential. J R Soc Interface. 2017 Dec;14(137):20170585. doi: 10.1098/rsif.2017.0585. PMID 29212756
- [Background] Hashish I, Haia HK, Harvey W, Feinmann C, Harris M. Reduction of postoperative pain and swelling by ultrasound treatment: a placebo effect. Pain. 1988 Jun;33(3):303-311. doi: 10.1016/0304-3959(88)90289-8. PMID 3419838
- [Background] Vase L, Robinson ME, Verne GN, Price DD. The contributions of suggestion, desire, and expectation to placebo effects in irritable bowel syndrome patients. An empirical investigation. Pain. 2003 Sep;105(1-2):17-25. doi: 10.1016/s0304-3959(03)00073-3. PMID 14499416